CLINICAL TRIAL: NCT07356128
Title: Binaural Cue Sensitivity in Children and Adults With Combined Electric and Acoustic Stimulation
Status: Recruiting | Type: Observational
Sponsor: Hearts for Hearing (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01DC020194 (NIH); 5R01DC020194 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Bilateral Sensorineural Hearing Loss; Cochlear Implant; Hearing Preservation; Electric and Acoustic Simulation
Keywords: sensorineural hearing loss; cochlear implant; electric and acoustic stimulation (EAS); hearing preservation
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children with normal hearing
  Interventions: Behavioral: binaural processing over time; Behavioral: binaural processing over time for children and adults with normal hearing
- Adults with normal hearing
  Interventions: Behavioral: binaural processing over time for children and adults with normal hearing
- Children with bilateral steeply sloping sensorineural hearing loss
  Interventions: Behavioral: binaural processing over time
- Adults with bilateral steeply sloping sensorineural hearing loss
  Interventions: Behavioral: binaural processing over time

INTERVENTIONS:
Behavioral: binaural processing over time — This study will not provide an intervention, but will study the effects of hearing technology on binaural processing for adults and children with bilateral steeply sloping sensorineural hearing loss
  Other Names: binaural development
  Groups: Adults with bilateral steeply sloping sensorineural hearing loss; Children with bilateral steeply sloping sensorineural hearing loss; Children with normal hearing
Behavioral: binaural processing over time for children and adults with normal hearing — Adults and children with normal hearing will be studied over time to characterize binaural processing and associated effects on speech perception in complex listening scenarios and spatial hearing abilities.
  Groups: Adults with normal hearing; Children with normal hearing

SUMMARY:
There is a rapidly growing population of adult and pediatric cochlear implant (CI) recipients with acoustic hearing preservation in the implanted ear(s) allowing for combined Electric and binaural Acoustic Stimulation (EAS). Despite the rapid technological and surgical advancements that have led to this increased prevalence, there is limited research on EAS outcomes-particularly for pediatric EAS listeners-including the expected trajectory of benefit following EAS fitting and underlying mechanisms driving benefit in EAS users of all ages. Thus, the purpose of this project is to provide a comprehensive description of behavioral and electrophysiologic measures of binaural hearing in adults and children both with normal hearing and EAS users.

DETAILED DESCRIPTION:
Cochlear implantation with minimally traumatic surgical techniques and atraumatic electrode arrays has led to an increasing prevalence of adult and pediatric cochlear implant (CI) recipients with the potential for combined Electric and binaural Acoustic Stimulation (EAS). Many studies have demonstrated that adult EAS users consistently exhibit significant benefits for speech understanding in noise and spatial hearing tasks as compared to a CI paired only with a contralateral HA. We have also demonstrated that sensitivity to interaural time difference (ITD) and interaural level difference (ILD) cues is correlated with EAS benefit for postlingually deafened adult listeners. Despite this active phase of discovery, there is still a striking paucity of research on EAS outcomes in pediatric CI users, the expected trajectory of benefit following EAS fitting, as well as underlying mechanisms driving EAS benefit (or lack thereof) in all populations. There is a disconnect between EAS availability and EAS utilization in all CI recipients and current audiological management of EAS candidates is not data driven. This is problematic given the protracted maturation of the binaural system and the fact that we do not understand what additional effects sensorineural hearing loss and combined EAS may have on the developing binaural system. The proposed research activities will describe the time course of binaural development using behavioral and objective responses to interaural differences in timing (phase) and level as well as allow for a natural factor investigation of a clinical intervention, the EAS fitting, on said development. Within the context of a clinical trial, we will compare acute and chronic EAS outcomes for speech recognition and spatial hearing as related to binaural cue sensitivity, cue weighting, and underlying neural synchrony necessary for ITD resolution. We have proposed a single-group assignment for both adult and pediatric EAS users and will also include chronological- and hearing-age-matched listeners with normal hearing (NH). A within-subjects, accelerated longitudinal design for both EAS and NH listeners will provide insight into the developmental trajectory of the binaural system for children NH and will provide a benchmark for interpreting effects of sensorineural hearing loss, asymmetry in audibility resulting from cochlear implantation, and EAS use on said trajectory. Our proposed research activities will help close the gap between what is technologically possible with EAS technology and what is clinically implemented by otologists and audiologists investigating development of binaural sensitivity and spatial hearing abilities. The resultant data will comprise the first comprehensive description of behavioral and electrophysiologic measures of binaural hearing in adults and children both with NH and EAS and will uncover information about our EAS clinical populations holding high potential for clinical application in device fittings as well as audiologic and otologic clinical recommendations regarding cochlear implantation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric EAS: aged 5-17; Adult EAS: aged 18+ years
* At least one CI and bilateral mild to profound sensorineural hearing loss with unaided audiometric thresholds ≤ 80 dB HL at 125 and 250 Hz, in both ears.

  * Willingness to use EAS technology in the implanted ear(s) to be verified via data logging
  * Nonverbal cognitive abilities within the typical range
  * No co-morbid diagnoses such as autism, auditory neuropathy, neurological disorder, or general cognitive impairment
  * Use of spoken English as main mode of communication
* For children and adults with normal hearing, they will demonstrate audiometric thresholds 20 dB HL or better from 250-8000 Hz

Exclusion Criteria:

* single-sided deafness (SSD)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with steeply sloping sensorineural hearing loss in both ears
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
EAS benefit for speech recognition in noise and spatial hearing abilities | 2 years
  For children and adults who are pursuing cochlear implantation with acoustic hearing preservation, we will describe the rate of hearing preservation following implantation. This is critical as it is well-known that individuals with acoustic hearing preservation achieve significantly higher scores on tasks of speech recognition in noise, particularly with diffuse noise.
Binaural cue sensitivity (interaural time and level differences) | 2 years
  For children and adults with precipitously sloping, high-frequency sensorineural hearing loss pursuing cochlear implantation, we will describe binaural cue sensitivity pre- and post-implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Hearts for Hearing, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the study is complete, we will make the fully de-identified data set available to investigators upon request.
Supporting Information: Study Protocol, ICF
Time Frame: November 30, 2028 is the anticipated date the de-identified IPD will be available. There is no end date determined as of yet.
Access Criteria: Interested investigators may reach out to the study PI (Rene Gifford, PhD) at rene.gifford@heartsforhearing.org to inquire about obtaining de-identified IPD starting November 30, 2028.

REFERENCES:
- [Background] Gifford RH, Dorman MF, Skarzynski H, Lorens A, Polak M, Driscoll CL, Roland P, Buchman CA. Cochlear implantation with hearing preservation yields significant benefit for speech recognition in complex listening environments. Ear Hear. 2013 Jul-Aug;34(4):413-25. doi: 10.1097/AUD.0b013e31827e8163. PMID 23446225
- [Background] Gifford RH, Davis TJ, Sunderhaus LW, Menapace C, Buck B, Crosson J, O'Neill L, Beiter A, Segel P. Combined Electric and Acoustic Stimulation With Hearing Preservation: Effect of Cochlear Implant Low-Frequency Cutoff on Speech Understanding and Perceived Listening Difficulty. Ear Hear. 2017 Sep/Oct;38(5):539-553. doi: 10.1097/AUD.0000000000000418. PMID 28301392
- [Background] Gifford RH, Stecker GC. Binaural cue sensitivity in cochlear implant recipients with acoustic hearing preservation. Hear Res. 2020 May;390:107929. doi: 10.1016/j.heares.2020.107929. Epub 2020 Feb 26. PMID 32182551
- [Background] Holder JT, Morrel W, Rivas A, Labadie RF, Gifford RH. Cochlear Implantation and Electric Acoustic Stimulation in Children With TMPRSS3 Genetic Mutation. Otol Neurotol. 2021 Mar 1;42(3):396-401. doi: 10.1097/MAO.0000000000002943. PMID 33555745
- [Background] Roberts JB, Stecker GC, Holder JT, Gifford RH. Combined Electric and Acoustic Stimulation (EAS) in Children: Investigating Benefit Afforded by Bilateral Versus Unilateral Acoustic Hearing. Otol Neurotol. 2021 Aug 1;42(7):e836-e843. doi: 10.1097/MAO.0000000000003139. PMID 33859136
- [Background] Gifford RH, Sunderhaus LW, Dawant BM, Labadie RF, Noble JH. Cochlear implant spectral bandwidth for optimizing electric and acoustic stimulation (EAS). Hear Res. 2022 Dec;426:108584. doi: 10.1016/j.heares.2022.108584. Epub 2022 Jul 28. PMID 35985964
- [Background] Reinhart P, Parkinson A, Gifford RH. Hybrid Cochlear Implant Outcomes and Improving Outcomes With Electric-Acoustic Stimulation. Otol Neurotol. 2024 Dec 1;45(10):e749-e755. doi: 10.1097/MAO.0000000000004305. PMID 39514431
- [Result] Fan Y, Gifford RH. Objective measure of binaural processing: Acoustic change complex in response to interaural phase differences. Hear Res. 2024 Jul;448:109020. doi: 10.1016/j.heares.2024.109020. Epub 2024 Apr 28. PMID 38763034

DOCUMENTS (2):
  • Informed Consent Form: Pediatric study participants (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT07356128/ICF_000.pdf
  • Informed Consent Form: Adult participants (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT07356128/ICF_001.pdf